CLINICAL TRIAL: NCT03841513
Title: Minimally Invasive Burch Colposuspension to Reduce Occult Stress Incontinence
Acronym: MICRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Friends of Prentice (Other)
Responsible Party: Principal Investigator, Sarah Collins, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00208016
Record Dates: First submitted 2019-01-23; First posted 2019-02-15 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence,Stress; Urinary Incontinence, Urge; Bowel Dysfunction; Sexual Dysfunction
Keywords: Burch Colposuspension; Sacrocolpopexy; Laparoscopy; Robotic Surgery
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress; Urinary Incontinence, Urge; Intestinal Diseases; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be assigned to one of two treatment groups with equal probability. A randomly permuted blocked randomization schema will be generated and maintained by a statistician not otherwise involved in the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study surgeons will provide clinical care to study participants, and therefore blinding the surgeon to treatment allocation is not feasible. However, we intend that all outcomes assessors and participants will be blinded to treatment allocation until 3-months outcomes are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in this arm will undergo standard laparoscopic or robotic sacrocolpopexy, without the addition of a laparoscopic/robotic Burch colposuspension
- Laparoscopic Burch Colposuspension (Active Comparator): Patients in this arm will undergo standard laparoscopic or robotic sacrocolpopexy, with the addition of a laparoscopic/robotic Burch colposuspension
  Interventions: Procedure: Laparoscopic Burch Colposuspension

INTERVENTIONS:
Procedure: Laparoscopic Burch Colposuspension — The Burch Colposuspension is an anti-incontinence procedure where non-absorbable monofilament suture is used in the retropubic space to form a suture bridge between the anterior vagina and Cooper's ligament, thereby gently elevating the anterior vaginal wall and providing urethral support.
  Arms: Laparoscopic Burch Colposuspension

SUMMARY:
This study evaluates the addition of a laparoscopic Burch colposuspension procedure at the time of laparoscopic sacrocolpopexy to prevent stress urinary incontinence. Half of the participants will undergo Burch colposuspension procedure at the time of sacrocolpopexy, and half of the participants will undergo sacrocolpopexy alone.

DETAILED DESCRIPTION:
In the United States it is estimated that 13% of women will undergo surgery for POP by age 80. In patients without symptoms of stress urinary incontinence (SUI), surgical correction of pelvic organ prolapse (POP) by itself can result in postoperative occult SUI. Two multicenter randomized trials of stress-continent women undergoing vaginal or open prolapse surgery showed lower rates of postoperative SUI if patients undergo concomitant anti-incontinence procedures. However, adverse outcomes vary based on the type of anti-incontinence procedure (open Burch colposuspension or retropubic midurethral sling) and route of surgery (open or vaginal), and therefore the preferred approach to address occult SUI is unknown.

Sacrocolpopexy is the gold standard surgical repair of pelvic organ prolapse of the apical compartment. The Burch colposuspension is a retropubic procedure in which the periurethral tissue of the anterior vagina is affixed to Cooper's ligament on either side using permanent suture bridges. In the Colpopexy and Urinary Reduction Efforts (CARE) trial patients without preoperative symptoms of SUI were randomized to receive or not to receive concomitant prophylactic Burch colposuspension at the time of abdominal sacrocolpopexy. At three months, the subjects who underwent the Burch procedure were found to have lower rates of SUI after surgery (33.6%) compared to the control group (57.4%). Furthermore, of patients who tested negative for SUI on preoperative urodynamic testing, 22.9 % of those who underwent the Burch procedure had SUI compared to 47.9% in the control group. Burch colposuspension did not increase the rate of urinary retention, urge incontinence, urinary urgency, urinary tract infection, intra or post-operative complications. The data in this trial supported the placement of prophylactic Burch colposuspension at the time of abdominal sacrocolpopexy.

Over the last decade, there has been a shift away from open routes of surgical access secondary to decreased morbidity and quicker recovery associated with minimally invasive procedures. As a result, open abdominal sacrocolpopexy with Burch colposuspension has fallen out of favor, and minimally invasive laparoscopic sacrocolpopexy is performed with greater frequency. Additionally, midurethral slings (MUS) have become the gold standard surgical procedure for the treatment of SUI and are performed more frequently than Burch colposuspension at the time of prolapse surgery. The Outcomes Following Vaginal Prolapse Repair and Midurethral Sling (OPUS) study examined the placement of prophylactic MUS at the time of vaginal prolapse surgery. Patients with MUS had lower rates of SUI than control group at 3 months (23.6% vs 49.4%) and at 12 months (27.3% vs 43%). However, unlike the CARE trial, patients with concomitant anti-incontinence procedure had higher rates of adverse events including bladder perforation (6.7% vs 0%), UTI (31.0% vs 18.3%), major bleeding (3.1% vs 0%), and incomplete bladder emptying at 6 weeks (3.7% vs 0%). In addition, MUS carries the risk of mesh erosion into the vagina or urinary tract.

By studying the addition of laparoscopic (including robotic) Burch colposuspension to laparoscopic sacrocolpopexy, the investigators anticipate optimizing surgical outcomes and minimizing complications for patients.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking and reading
* Symptomatic pelvic organ prolapse with any compartment at or beyond the hymen
* Stress-continent, as defined as response of "no" to question 17 of PFDI-20: "Do you usually experience urine leakage related to coughing, sneezing, or laughing?", as well as a negative empty supine stress test.
* Planning laparoscopic or robotic sacrocolpopexy, with or without hysterectomy
* Have completed childbearing

Exclusion Criteria:

* Adults unable to consent
* Pregnant women or patients desiring future pregnancy
* Patients undergoing uterine sparing surgery
* Individuals under age 18
* Prior procedure for stress urinary incontinence
* Prior retropubic surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Collins, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University Prentice Women's Hospital, Chicago, Illinois
  - Loyola University Hospital, Maywood, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu JM, Matthews CA, Conover MM, Pate V, Jonsson Funk M. Lifetime risk of stress urinary incontinence or pelvic organ prolapse surgery. Obstet Gynecol. 2014 Jun;123(6):1201-1206. doi: 10.1097/AOG.0000000000000286. PMID 24807341
- [Background] Brubaker L, Cundiff GW, Fine P, Nygaard I, Richter HE, Visco AG, Zyczynski H, Brown MB, Weber AM; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy with Burch colposuspension to reduce urinary stress incontinence. N Engl J Med. 2006 Apr 13;354(15):1557-66. doi: 10.1056/NEJMoa054208. PMID 16611949
- [Background] Wei JT, Nygaard I, Richter HE, Nager CW, Barber MD, Kenton K, Amundsen CL, Schaffer J, Meikle SF, Spino C; Pelvic Floor Disorders Network. A midurethral sling to reduce incontinence after vaginal prolapse repair. N Engl J Med. 2012 Jun 21;366(25):2358-67. doi: 10.1056/NEJMoa1111967. PMID 22716974
- [Background] Geller EJ, Siddiqui NY, Wu JM, Visco AG. Short-term outcomes of robotic sacrocolpopexy compared with abdominal sacrocolpopexy. Obstet Gynecol. 2008 Dec;112(6):1201-1206. doi: 10.1097/AOG.0b013e31818ce394. PMID 19037026
- [Background] Hsiao KC, Latchamsetty K, Govier FE, Kozlowski P, Kobashi KC. Comparison of laparoscopic and abdominal sacrocolpopexy for the treatment of vaginal vault prolapse. J Endourol. 2007 Aug;21(8):926-30. doi: 10.1089/end.2006.0381. PMID 17867956
- [Background] Paraiso MF, Walters MD, Rackley RR, Melek S, Hugney C. Laparoscopic and abdominal sacral colpopexies: a comparative cohort study. Am J Obstet Gynecol. 2005 May;192(5):1752-8. doi: 10.1016/j.ajog.2004.11.051. PMID 15902189

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Laparoscopic Burch Colposuspension
Started | 24 | 26
Completed | 24 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Laparoscopic Burch Colposuspension | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Full Range); unit: years] | 61 [52 to 69] | 66 [61 to 69] | 64 [52 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 22 | 24 | 46
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
BMI [Mean (Inter-Quartile Range); unit: kg/m^2] | 25.1 [22.4 to 30.7] | 25.6 [24.0 to 26.8] | 25.4 [23.2 to 28.8]
Baseline POP-Q Stage [Median (Inter-Quartile Range); unit: stage] — The plane of the hymen being defined as zero, all measures are in centimeters above / proximal to the hymen. Once all measurements have been made the stage of the prolapse can be identified; Stage 0: No prolapse is observed. Stage 1: The most proximal portion of prolapse is greater than 1 cm above the level of the hymen. Stage 2: The most proximal portion of prolapse is found between 1 cm higher than hymen and 1cm beneath hymen. Stage 3: The most distal part of the prolapse extends more than 1cm beneath the hymen but no further than 2 cm. Stage 4: vaginal eversion has taken place.
  stage | 3 [3 to 3] | 3 [3 to 3] | 3 [3 to 3]
POPDI [Mean (Standard Deviation); unit: scores on a scale] — Pelvic Organ Prolapse Distress Inventory. To provide a symptom inventory and to measure the degree of bother and distress caused by the broad array of pelvic floor symptoms, in particular related to pelvic organ prolapse. The responses are scored to generate a total POPDI-6 score, which can range from 0 to 100, with higher scores indicating greater distress.
  scores on a scale | 47.7 (23.0) | 35.7 (24.3) | 41.7 (23.6)
CRADI [Median (Full Range); unit: score on a scale] — he Colorectal Anal Distress Inventory (CRADI) is a questionnaire used to assess the level of distress experienced by individuals with bowel symptoms. The CRADI score is calculated by taking the mean value of all answered questions and then multiplying by 25 (range 0 to 100). Higher score means worse symptom and distress.
  score on a scale | 23.4 [7.0 to 39.1] | 14.1 [6.3 to 41.4] | 18.8 [6.3 to 41.4]
UDI [Median (Full Range); unit: score on a scale] — The Urinary Distress Inventory (UDI) is a questionnaire used to assess the impact of urinary symptoms on a person's life. It helps measure the severity of symptoms like frequent urination, urine leakage, and voiding difficulties, as well as how much these symptoms bother the individual. It's scored by summing the responses to 6 questions, each with a rating scale of 0-3 (not at all to greatly). A higher total score indicates greater distress and impact on quality of life. The final score is then adjusted to a 0-100 scale.
  score on a scale | 22.9 [8.3 to 36.5] | 25.0 [7.3 to 38.5] | 24.0 [7.3 to 38.5]
PISQ-12 [Mean (Standard Deviation); unit: score on a scale] — PISQ-12 (Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire, 12-item form), each of the 12 questions is scored on a Likert scale from 0 (always) to 4 (never). Items 1-4 are reverse-scored, meaning "always" is scored as 4 and "never" as 0, and the reverse for items 5-12. The total score is the sum of all 12 item scores, ranging from 0 to 48. A higher score indicates better sexual function.
  score on a scale | 13.8 (5.8) | 15.1 (6.2) | 14.5 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stress Urinary Incontinence
Description: Rate of Stress Urinary Incontinence, as defined as a participant satisfying one or more of the following:
  * A positive retro-fill cough stress test at 300mL
  * Answer of "yes" to question #17 of Pelvic Floor Distress Inventory 20 (PFDI-20)
  * Any treatment for stress urinary incontinence after the study surgery
Time Frame: 3 months following study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Laparoscopic Burch Colposuspension
Number analyzed (Participants) | 24 | 26
Participants | 10 | 13

2. Secondary Outcome: Number of Participants With Urinary Urgency Incontinence
Description: Rate of Urgency Urinary Incontinence, as defined as a participant satisfying one or more of the following:
  * Answer of "yes" to question #16 of Pelvic Floor Distress Inventory 20 (PFDI-20)
  * Any treatment for urgency urinary incontinence after the study surgery
Time Frame: 3 months following study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Laparoscopic Burch Colposuspension
Number analyzed (Participants) | 24 | 26
Participants | 1 | 2

3. Secondary Outcome: Number of Participate With Urinary Frequency
Description: Values based on response of "moderately" or "quite a bit" to Question #15 of PFDI-20: "Do you usually experience frequent urination?"
Time Frame: 3 months following study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Laparoscopic Burch Colposuspension
Number analyzed (Participants) | 24 | 26
Participants | 2 | 4

4. Secondary Outcome: Number of Participants With Urinary Retention
Description: Rate of Urinary Retention, defined as a post void residual greater than 150 mL obtained via straight catheterization
Time Frame: 3 months following study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Laparoscopic Burch Colposuspension
Number analyzed (Participants) | 24 | 26
Participants | 1 | 3

5. Secondary Outcome: Number of Participants With Urinary Tract Infection
Description: Rate of Urinary Tract Infection, defined as a positive urine culture obtained from a straight catheterized urine specimen, from participants with symptoms of urinary tract infection (fever, dysuria, urinary urgency, urinary frequency).
Time Frame: 3 months following study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Laparoscopic Burch Colposuspension
Number analyzed (Participants) | 24 | 26
Participants | 2 | 1

6. Secondary Outcome: Pelvic Organ Prolapse Symptoms
Description: Compare Pelvic Organ Prolapse Symptoms utilizing the Pelvic Floor Distress Inventory 20 (PFDI-20), questions #1-6. Participants respond to each question on a scale of 0 to 4, with higher scores indicating greater dysfunction. The sum of scores is reported for this subscale, with a minimum score of 0 and maximum score of 24.
Time Frame: 3 months following study intervention
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control | Laparoscopic Burch Colposuspension
Number analyzed (Participants) | 24 | 26
score on a scale | 8.3 [0 to 11.9] | 2.1 [0 to 12.5]

7. Secondary Outcome: Bowel Symptoms
Description: Compare Bowel Symptoms utilizing the Pelvic Floor Distress Inventory 20 (PFDI-20), questions #7-14. Participants respond to each question on a scale of 0 to 4, with higher scores indicating greater dysfunction. The sum of scores is reported for this subscale, with a minimum score of 0 and maximum score of 32.
Time Frame: 3 months following study intervention
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control | Laparoscopic Burch Colposuspension
Number analyzed (Participants) | 24 | 26
score on a scale | 6.3 [0 to 17.2] | 6.7 [0 to 24.2]

8. Secondary Outcome: Sexual Function
Description: Compare Sexual Function utilizing the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire 12 (PISQ-12). Participants respond to each question on a scale of 0 to 4, with higher scores indicating greater dysfunction. The sum of scores is reported for this subscale, with a minimum score of 0 and maximum score of 48.
Time Frame: 3 months following study intervention
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control | Laparoscopic Burch Colposuspension
Number analyzed (Participants) | 24 | 26
score on a scale | 10.5 [8.8 to 15.2] | 12.0 [11.0 to 17.0]

9. Secondary Outcome: Number of Participants With Surgical Complication
Description: Compare rate of intraoperative and short-term surgical complications, as defined by the Dindo classification system.
Time Frame: 3 months following study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Laparoscopic Burch Colposuspension
Number analyzed (Participants) | 24 | 26
Participants | 3 | 5

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control | Laparoscopic Burch Colposuspension
All-Cause Mortality (participants affected / at risk) | 3/24 | 5/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT03841513/Prot_SAP_000.pdf